CLINICAL TRIAL: NCT02708173
Title: Safety Study of Quadrivalent Influenza Virus Vaccine in Healthy People Aged 3 Years and Older
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Chaoyang District Centre for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: cycdc2015-5
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-03

CONDITIONS: Quadrivalent Influenza Virus Vaccine
Keywords: vaccine; safety

ARMS (2):
- One dose Vaccine in aged 18-60 years old (Experimental): One dose of Quadrivalent Influenza Virus Vaccine will be given in aged 18-60 years old.
  Interventions: Biological: One dose of Quadrivalent Influenza Virus Vaccine
- One dose Vaccine in aged 3-17 years old (Experimental): One dose of Quadrivalent Influenza Virus Vaccine will be given in aged 3-17 years old.
  Interventions: Biological: One dose of Quadrivalent Influenza Virus Vaccine

INTERVENTIONS:
Biological: One dose of Quadrivalent Influenza Virus Vaccine
  Arms: One dose Vaccine in aged 18-60 years old
Biological: One dose of Quadrivalent Influenza Virus Vaccine
  Arms: One dose Vaccine in aged 3-17 years old

SUMMARY:
This study evaluates the safety of Quadrivalent Influenza Virus Vaccine in Healthy People Aged years 3 to 60.40 Subjects will be equally divided into 2 groups,including 3-17 years old and 18-60 years old.Adult group first receive one dose of Quadrivalent Influenza Virus Vaccine.Then minors group also receive one dose of Quadrivalent Influenza Virus Vaccine after 7 days.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects more than 3 years old, and the subjects can be informed consent, and sign the informed consent.
* the subjects and his guardians can obey the demands of the scheme .
* Axillary temperature less than 37℃

Exclusion Criteria:

* The people who has a vaccine allergies, or who allergic to any kind of composition in experimental vaccine, such as eggs,ovalbumin etc.
* The people who has serious side effects to vaccine, such as allergy,urticaria, skin eczema, dyspnea, angioneurotic edema or abdominal pain.
* the subject who has symptoms of acute infection within a week.
* Autoimmune diseases or Immune function defect, people has immunosuppressive therapy, cytotoxic treatment or inhaled corticosteroids in the past 6 months.
* People has congenital malformations, developmental disorder or serious chronic diseases( such as Down's syndrome, diabetes, Sickle cell anemia or nerve system disease)
* People has asthma Unstable that need emergency treatment, hospitalization, intubation, oral or intravenous corticosteroid in the past 2 years.
* Diagnosed abnormal coagulation(Lack of clotting factors,Clotting disorders,Platelet abnormality) or significant bruising or coagulopathy
* people has history or family history of convulsions, seizures, encephalopathy and psychiatric.
* alienia, functional asplenia, and alienia or splenectomy in any situation.
* Serious neurological disorders such as Green Barry syndrome.
* people who has received blood products or immunoglobulin products in the past one months.
* people who has received other study drug in the past one month.
* people who received live attenuated vaccine, subunit vaccine or inactivated vaccine.
* people who has received allergy treatment in in the past 14 days.
* People who is on anti-TB treatment.
* People whose axillary temperature is more than 37℃ before the vaccination.
* People who is pregnant.
* Any factors unsuitable for clinical trail according to the researchers.

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The rate of adverse reactions of Quadrivalent Influenza Virus Vaccine | 3 months
  Adverse reactions associated with vaccine will be observed in subjects after vaccination. Solicited local adverse events include Pain, Redness, Swelling, Induration, Rash, Pruritus at injection site. solicited general adverse events include Fever, Nausea, Vomiting, Diarrhea, Decreased appetite, Be agitated (irritability, abnormal crying), fatigue, allergy

CONTACTS AND LOCATIONS:
Locations (1):
- DongBa clinical center, Beijing, Beijing Municipality, China